CLINICAL TRIAL: NCT02880033
Title: Modulation of Oxidative Stress and Apoptosis of Energy Metabolism by Deferiprone From the Circulating Lymphocytes of Patients With Parkinson's Disease or Amyotrophic Lateral Sclerosis
Brief Title: Oxidative Stress and Apoptosis of Energy Metabolism by Deferiprone From the Circulating Lymphocytes
Acronym: LymphoEnergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010_29; 2010-A01216-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-03; First posted 2016-08-26 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Parkinson's Disease; Amyotrophic Lateral Sclerosis; Oxidative Stress; Iron Overload
Keywords: Parkinson's disease; Amyotrophic lateral sclerosis; Peripheral blood mononuclear cells; ex vivo model for oxidative stress; iron metabolism and chelation
MeSH Terms: conditions — Parkinson Disease; Amyotrophic Lateral Sclerosis; Iron Overload | interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Parkinson's disease (Active Comparator): ex vivo analysis of lymphocytes from 30 patients with Parkinson's disease with deferiprone and placebo treatment
  Interventions: Drug: deferiprone; Drug: placebo
- Amyotrophic lateral sclerosis (Active Comparator): ex vivo analysis of lymphocytes from 30 patients with Amyotrophic lateral sclerosis with deferiprone and placebo treatment
  Interventions: Drug: deferiprone; Drug: placebo
- healthy age and sex matched controls (Placebo Comparator): ex vivo analysis of lymphocytes from 30 healthy age and sex matched controls with deferiprone and placebo treatment
  Interventions: Drug: deferiprone; Drug: placebo

INTERVENTIONS:
Drug: deferiprone — to test the action of deferiprone on lymphocytes from patients and controls ex vivo
  Other Names: FERRIPROX
Drug: placebo — to control the action of placebo on lymphocytes from patients and controls ex vivo

SUMMARY:
Peripheral blood mononuclear cells (PBMC) and platelets could be interesting ex vivo models to study brain diseases. Indeed, there is no access to neurons from patients. However, PBMC can exhibit different physiopathological mechanisms that are ubiquitous (i.e. oxidative stress, mitochondriopathy with energy metabolism, inflammation, protein folding, iron metabolism and programmed cell death ...). The platelets are pivotal in the healing system with large range of growth factors. A new therapeutic concept of conservative iron chelation with deferiprone for neuroprotection is under development.

The action of deferiprone on the different mechanisms and notably the oxidative stress are to obtain from a collection of PBMC and platelets from patient having Parkinson's disease and Amyotrophic lateral sclerosis and healthy controls to study ex vivo.

PBMC and platelets will be stored for future analyses.

DETAILED DESCRIPTION:
The study collection of PBMC and platelets from 30 patient having Parkinson's disease 30 patients having Amyotrophic lateral sclerosis and 30 healthy controls.

The collection will be performed either by cytapheresis for half of the patient and by collecting the whole blood for the other half.

PBMC and platelets will be stored at minus 80°C. PBMC of patients and controls are exposed ex vivo to different pathological condition (mainly Hydrogen peroxide, menadione, hypoxia...) with and without deferiprone to analyse whether the level of oxidative stress (Reactive Oxygen Species and notably hydroxyl radical with hydroxypethidine probe with flow cytometry) is reduced under deferiprone (primary criterion. Secondary analyses will concern the level of iron, the energy metabolism (aerobic versus anaerobic and the level of Adenosine triphosphate production), the type of cell death (apoptosis, autophagy and new programmed cell death: Ferroptosis) and inflammation. Finally, the level of growth factors and their effectiveness will be studied from platelets.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease according to Movement Disorders Society criteria
* Amyotrophic Lateral Sclerosis according to El escorial criteria
* Age and sex matched healthy controls

Exclusion Criteria:

* Severe comorbidities (cancer, other degenerative diseases, hemopathy, inflammatory diseases)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2019-10 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
hydroxyl radical measured | 12 months
  hydroxypethidine probe with Fluorescence-activated cell sorting

SECONDARY OUTCOMES:
adenosine triphosphate production measured by seahorse | 12 months
  seahorse experimentation
oxygen consumption measured by seahorse | 12 months
  seahorse experimentation
free reactive iron (ferrous iron) | 12 months
  calceine assay
lipid peroxidation measured by Fluorescence-activated cell sorting | 12 months
  flow cytometry with bodipy probe

CONTACTS AND LOCATIONS:
Overall Officials: David DEVOS, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No